CLINICAL TRIAL: NCT02010697
Title: Mail Campaigns That Target Smokers or Nonsmokers Who Live With Smokers
Brief Title: Nonsmokers Helping Smokers Quit
Acronym: Project BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UO1 CA154280 IRB #130764; U01CA154280 (NIH)
Record Dates: First submitted 2013-12-02; First posted 2013-12-13 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; nonsmokers; proxy; mail intervention; self-help; behavioral intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Messages targeting nonsmokers (Experimental): Messages targeting nonsmokers include 10 mailings for nonsmokers sent over 10 weeks. The mailed materials include postcards, informational materials, CDs, DVDs, coupons for cessation-related incentives such as nicotine patches, and links to secured websites. The mail campaign is augmented with brief phone calls to ensure receipt of mailings and to reinforce targeted messages.
  Interventions: Behavioral: Messages targeting nonsmokers
- Messages targeting smokers (Experimental): Messages targeting smokers include 10 mailings for smokers sent over 10 weeks. The mailed materials include postcards, informational materials, CDs, DVDs, coupons for cessation-related incentives such as nicotine patches, and links to secured websites. The mail campaign is augmented with brief phone calls to ensure receipt of mailings and to reinforce targeted messages.
  Interventions: Behavioral: Messages targeting smokers
- Usual care (No Intervention): one time mailing with a self-help quit kit

INTERVENTIONS:
Behavioral: Messages targeting nonsmokers
  Arms: Messages targeting nonsmokers
Behavioral: Messages targeting smokers
  Arms: Messages targeting smokers

SUMMARY:
This study examines whether nonsmokers can be mobilized to help smokers quit. We will test, via mail campaign, whether targeting nonsmokers can be equally effective in increasing smokers' quit rate as targeting smokers directly. The hypothesis is that both targeted interventions will lead to a higher quit rate than a control group, which receives one set of self-help materials. Each of the targeted intervention groups receives 10 mailings. Smoking status of all three groups will be measured at 3 and 7 months post randomization.

DETAILED DESCRIPTION:
This study examines the potential of enlisting nonsmokers to help smokers quit smoking. Nonsmokers are the majority of the society. If an intervention can be designed to mobilize nonsmokers to help smokers quit, then it has strong implications for increasing smoking cessation at the population level. The conventional approach in smoking cessation is to target smokers directly. This study aims to test whether targeting nonsmokers can be equally effective. The study employs a three arm randomized design, in which a smoker-nonsmoker pair in the same household will be randomized into one of the three groups. One group receives materials targeting the smoker in the household, one group receives materials targeting the nonsmoker, and the third group serve as a control group. The intervention consists of mailed materials which include postcards, informational materials, CDs, DVDs, coupons for cessation-related incentives such as nicotine patches, and links to secured websites. The mail campaign is augmented with brief phone calls to ensure receipt of mailings and to reinforce targeted messages.The mail campaign is augmented with brief phone calls to ensure receipt of mailings and to reinforce targeted messages. At 3 and 7 months post randomization, project staff contact all participants to assess their smoking status.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* A household with at least one smoker and one nonsmoker
* Valid contact information
* English proficiency, both speaking and reading

Exclusion Criteria:

* Insufficient contact information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3125 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Messages Targeting Nonsmokers: Messages targeting nonsmokers include 10 mailings for nonsmokers sent over 10 weeks. The mailed materials include postcards, informational materials, CDs, DVDs, coupons for cessation-related incentives such as nicotine patches, and links to secured websites. The mail campaign is augmented with brief phone calls to ensure receipt of mailings and to reinforce targeted messages.
  Messages targeting nonsmokers
- Messages Targeting Smokers: Messages targeting smokers include 10 mailings for smokers sent over 10 weeks. The mailed materials include postcards, informational materials, CDs, DVDs, coupons for cessation-related incentives such as nicotine patches, and links to secured websites. The mail campaign is augmented with brief phone calls to ensure receipt of mailings and to reinforce targeted messages.
  Messages targeting smokers
Period: Overall Study
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care
Started | 1044 | 1038 | 1043
Completed | 1044 | 1038 | 1043
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care | Total
Number analyzed (Participants) | 1044 | 1038 | 1043 | 3125
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 116 | 91 | 109 | 316
  25-44 | 487 | 479 | 496 | 1462
  45-64 | 409 | 420 | 408 | 1237
  65+ | 32 | 48 | 30 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 566 | 590 | 566 | 1722
  Male | 478 | 448 | 477 | 1403
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 491 | 481 | 542 | 1514
  Black | 289 | 310 | 275 | 874
  Hispanic | 121 | 107 | 88 | 316
  Asian | 9 | 9 | 11 | 29
  AIAN | 61 | 46 | 61 | 168
  Multi | 73 | 85 | 65 | 223
  Other | 0 | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  0 to 8 | 40 | 45 | 40 | 125
  9 to 12 | 231 | 202 | 228 | 661
  HSD/GED | 343 | 338 | 335 | 1016
  Some College | 372 | 381 | 391 | 1144
  BS+ | 58 | 72 | 49 | 179

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting 30-day Abstinence
Description: Assessment interview is conducted over the phone at 7-months post enrollment to determine 30-day abstinence. The interview will cover, as appropriate, tobacco use, use of quitting aids, and pattern of quitting (including slips and relapse situations).
Time Frame: 7-months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care
Number analyzed (Participants) | 1044 | 1038 | 1043
Participants | 203 | 222 | 135

2. Secondary Outcome: Support for Quitting
Description: The number of participants who felt they had "a lot" of support for quitting or staying quit.
Time Frame: At intake
Measure: Count of Participants; unit: Participants
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care
Number analyzed (Participants) | 1044 | 1038 | 1043
Participants | 690 | 712 | 704

3. Secondary Outcome: Number of Participants Reporting 30-day Abstinence
Description: Assessment interview is conducted over the phone at 3-months post enrollment to determine 30-day abstinence. The interview will cover, as appropriate, tobacco use, use of quitting aids, and pattern of quitting (including slips and relapse situations).
Time Frame: 3-months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care
Number analyzed (Participants) | 1044 | 1038 | 1043
Participants | 120 | 137 | 56

4. Other Pre Specified Outcome: Counseling
Description: Did participants receive counseling
Time Frame: 7-months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care
Number analyzed (Participants) | 1044 | 1038 | 1043
Participants | 20 | 58 | 0

ADVERSE EVENTS:
Arm/Group | Messages Targeting Nonsmokers | Messages Targeting Smokers | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/1044 | 0/1038 | 0/1043
Other Adverse Events (participants affected / at risk) | 0/1044 | 0/1038 | 0/1043

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No